CLINICAL TRIAL: NCT06033274
Title: Global Multicenter Registry on Transcatheter TRIcuspid Valve RePLACEment: the TRIPLACE Registry
Brief Title: Global Multicenter Registry on Transcatheter TRIcuspid Valve RePLACEment
Acronym: TRIPLACE
Status: Recruiting | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: The Cleveland Clinic (Other); University of Toronto (Other); University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-15312
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Tricuspid Regurgitation
Keywords: valvular heart disease; tricuspid regurgitation; transcatheter tricuspid valve replacement
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Tricuspid Regurgitation undergoing Transcatheter Tricuspid Valve Replacement: Patients having clinically significant tricuspid regurgitation, defined according to current guidelines (ESC/EACTS and ACC/AHA) for valvular heart disease, requiring transcatheter tricuspid valve replacement
  Interventions: Device: Transcatheter Tricuspid Valve Replacement

INTERVENTIONS:
Device: Transcatheter Tricuspid Valve Replacement — All patients undergoing Transcatheter Tricuspid Valve Replacement for native tricuspid valve disease

SUMMARY:
The field of transcatheter tricuspid valve replacement (TTVR) is rapidly emerging and data on this topic are scarce. Particularly, little is known about which patients are at greatest risk of procedural complications, such as the timing and onset of conduction disturbances necessitating permanent pacemaker implantation, and how such patients are managed. On this background, the TRIPLACE Registry - an investigator-initiated global multicenter registry - is aimed at better understanding the safety and efficacy of orthotopic TTVR.

DETAILED DESCRIPTION:
The primary aims of the registry will be:

* To examine the safety, efficacy, and long-term outcomes of TTVR
* To assess the incidence of procedural complications and their correlations with adverse clinical outcomes
* To investigate the impact of different pre/post-procedural factors on peri-procedural complications and long-term outcomes after TTVR
* To explore the characteristics of patients deemed eligible for TTVR.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Transcatheter Tricuspid Valve Replacement
* Native Tricuspid Valve disease
* Orthotopic Tricuspid Valve Implantation

Exclusion Criteria:

* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing orthotopic Transcatheter Tricuspid Valve Replacement for clinically significant tricuspid valve disease.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Freedom from device-related complications | 30 days after the index procedure
  Freedom from device-related complications will be determined by assessing the number of participants with procedural, peri-procedural and device-related complications
Reduction in Tricuspid Regurgitation Severity | 30 days after the index procedure
  Tricuspid Regurgitation measured by transthoracic echocardiography. Assessment of MI severity according to current guidelines (ESC/EACTS and ACC/AHA) for valvular heart disease.
  Tricuspid Regurgitation is measured by transthoracic echocardiography in accordance with current guidelines (ESC/EACTS and ACC/AHA) for valvular heart disease. Mean tricuspid regurgitation severity will be determined using the following scale: 0=none/trace; 1=mild; 2=moderate; 3=severe; 4=massive; 5=torrential. Change from baseline tricuspid regurgitation severity score 30 days after baseline will be assessed

SECONDARY OUTCOMES:
Permanent Pacemaker Implantation | 30 days after the index procedure
  The number of participants who have received a permanent pacemaker implantation will be recorded
Combined all-cause mortality or rehospitalization for congestive heart failure | 12 months after the index procedure
  The composite of mortality from any cause and participants re-hospitalized for acute decompensated congestive heart failure will be recorded
All-cause mortality | 12 months after the index procedure
  The number of deaths due to any cause will be recorded
Hospitalization for congestive heart failure | 12 months after the index procedure
  The number of participants who have been hospitalized with acute decompensated congestive heart failure will be recorded
The number of participants with New York Heart Association (NYHA) Stage III or IV heart failure | 12 months after the index procedure
  The number of participants who meet either NYHA III or NYHA IV classifications for heart failure will be recorded.
  NYHA Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest
  NYHA Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients
Device Thrombosis | 12 months after the index procedure
  The number of participants who have been identified with device thrombosis will be recorded
Tricuspid Regurgitation Severity | 12 months after the index procedure
  Tricuspid Regurgitation is measured by transthoracic echocardiography. Assessment of MI severity will be conducted in accordance with current guidelines (ESC/EACTS and ACC/AHA) for valvular heart disease. Mean tricuspid regurgitation severity will be determined using the following scale: 0=none/trace; 1=mild; 2=moderate; 3=severe; 4=massive; 5=torrential. Higher mean scores are indicative of greater TR severity
Quality of Life - Kansas City Cardiomyopathy Questionnaire | 12 months after the index procedure
  Quality of Life is evaluated using the Kansas City Cardiomyopathy Questionnaire (KCCQ). The KCCQ has a 2-week recall period and includes 23 items that map to 7 domains: symptom frequency; symptom burden; symptom stability; physical limitations; social limitations; quality of life; and self-efficacy (the patient's understanding of how to manage their heart failure). The symptom frequency and symptom burden domains are merged into a total symptom score, which can be combined with the physical limitation domain to create a clinical summary score that mirrors the key concepts of the NYHA functional class. The symptom, physical limitations, social limitations, and quality of life domains are combined to create an overall summary score, which is the primary health status outcome All scores are represented on a 0-to-100-point scale, where lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life
Tricuspid Valve Reintervention | 12 months after the index procedure
  The number of participants who undergo tricuspid valve surgical and/or transcatheter reintervention will be summed and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scotti, MD, Principal Investigator — Montefiore Medical Center; Azeem Latib, MD, Principal Investigator — Montefiore Medical Center; Rishi Puri, MD, Principal Investigator — The Cleveland Clinic; Neil Fam, MD, Principal Investigator — St. Michaels Hospital; Thomas Modine, MD, Principal Investigator — University Hospital, Bordeaux
Locations (21):
- United States (5):
  - Arizona Heart Hospital (Biltmore Cardiology), Phoenix, Arizona
  - Columbia University Irving Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
- Canada (3):
  - St. Paul's Hospital, Vancouver, British Columbia
  - St Michael's Hospital, University of Toronto, Toronto, Ontario
  - Quebec Heart and Lung Institute, Laval University, Quebec City, Quebec, Canada, Québec, Quebec
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark
- France (3):
  - Chu De Bordeaux - Haut-Lévêque Hospital, Bordeaux, Pessac
  - Centre Hospitalier Universitaire de Lille, Lille
  - Clinique Pasteur Toulouse, Toulouse
- Germany (6):
  - Heart and Diabetes Centre, North Rhine-Westphalia (NRW), Ruhr-University, Bad Oeynhausen
  - Heart Center Cologne, University of Cologne, Cologne
  - Cardiovascular Center (CVC) Frankfurt, Division of Cardiology, Frankfurt
  - University Heart and Vascular Center, Department of Cardiology, Hamburg
  - University Heart Center, Schleswig-Holstein University, Lübeck
  - Medical Clinic and Polyclinic, University Hospital of Munich (LMU Klinikum), Munich
- Italy (2):
  - San Raffaele University Hospital, Milan
  - Centro Cardiologico Monzino IRCCS, Milan
- University Hospital Alvaro Cunqueiro (CHUVI), Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scotti A, Puri R, Sturla M, Zahr F, Boone R, Kodali S, Tchetche D, De Backer O, Coisne A, Ludwig S, Stolz L, Estevez Loureiro R, Adam M, De Marco F, Ho EC, Cheung A, Moey M, Ong G, Chadderdon S, Lulic D, Bartkowiak J, Echarte J, Sievert H, Byrne T, Maisano F, Frerker C, Dumonteil N, Oliva OA, Rudolph TK, Kirchner J, Bakhtadze B, Kapadia SR, Rodes-Cabau J, Schofer N, Granada J, Hausleiter J, Hahn RT, Modine T, Fam N, Latib A. Incidence, Predictors, and Management of Conduction Disturbances After Transcatheter Tricuspid Valve Replacement: The TRIPLACE Registry. JACC Cardiovasc Interv. 2025 Jul 28;18(14):1789-1799. doi: 10.1016/j.jcin.2025.05.029. Epub 2025 Jul 9. PMID 40637674
- [Derived] Traynor BP, Scotti A, Puri R, Sturla M, Zahr F, Boone R, Kodali S, Tchetche D, De Backer O, Coisne A, Ludwig S, Stolz L, Loureiro RE, Adam M, De Marco F, Biroli M, Ho EC, Cheung A, Patrascu A, Alnasser S, Chadderdon S, Lulic D, Bartkowiak J, Echarte-Morales J, Sievert H, Byrne T, Maisano F, Frerker C, Dumonteil N, Oliva OA, Rudolph TK, Rudolph F, Krishnaswamy A, Kapadia SR, Portillo JD, Rodes-Cabau J, Schofer N, Granada JF, Hausleiter J, Hahn RT, Modine T, Latib A, Fam N. Transcatheter Tricuspid Valve Replacement in Patients With Cardiac Implantable Electronic Device Leads: The TRIPLACE Registry. JACC Clin Electrophysiol. 2026 Jan 20:S2405-500X(25)01104-1. doi: 10.1016/j.jacep.2025.12.027. Online ahead of print. PMID 41575411